CLINICAL TRIAL: NCT04376099
Title: Focus Sur l'Analyse de la récupération en oxymétries transcutanées (French Language)
Brief Title: Focus on Analysis of Recovery in Oximetry
Acronym: FARO
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/42
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise oximetry: Patients complaining claudication and referred for exercise diagnostic oximetry. Exercise oximetry are performed on treadmill (3.2km/h, 10% slope)
  Interventions: Diagnostic Test: Transcutaneous oxygen pressure measurement during the treadmill test

INTERVENTIONS:
Diagnostic Test: Transcutaneous oxygen pressure measurement during the treadmill test — Calculation of the decrease from rest of oxygen pressure (DROP) throughout the period of rest exercise and recovery.
  The DROP is calculated as chanegs on each limb probe minus changes on a chest reference probe from rest.
  Analysis of the recovery period of the recordings will be done to seach for recovery 50% and 90% from the minimal DROP observed Evaluation of calf and non calf pain during the tests. Evaluation of calf and non calf (buttock or thigh) ischemia during the tests. Ischemia being defined as a monimal DROP lower than minus 15 mmHg.

SUMMARY:
Analysis of localizations for symptoms and ischemia on treadmill and of the recovery profiles of patients that have had an exercise oximetry

DETAILED DESCRIPTION:
Patients referred for exercise oximetry have buttocks thighs and calves recording during exercise and in the recovery period for a minimum of 10 minutes.

For each limb probe the decrease from rest of oxygen pressure (DROP) index is calculated as a subtraction of chest changes from limb changes throughout rest, exercise and recovery. DROP was measured as a routine on buttocks, thighs and calves and a minimal DROP lower than minus 15 mmHg considered indicative of the presence of regional blood flow impairment (ischemia) in the considered area.

Recordings and patients characteristics are recorded on a institutionally validated database.

A comparison will be performed of symptoms by history to symptoms reported on treadmill and hemodynamic results attained through DROP values.

Re-analysis of the recordings after ethical approval will be performed in an aim at estimating the duration of 50% and 90% recovery of DROP at the different levels (buttocks tigh and calves) to account for hemodynamic impairmenty not only at the calf (calves) level.

ELIGIBILITY:
Inclusion Criteria:

* Available exercise oximetry recording

Exclusion Criteria:

* Deny of the use of the medical file from the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred for exercise oximetry for intermittent claudication
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Transcutanesous oximetry DROP index 50% recovery time | Maximum 30 minutes (duration of the recovery phase)
  Time for the DROP index to reach 50% of its minimal value from the end of walking

SECONDARY OUTCOMES:
Transcutanesous oximetry DROP index 90% recovery time | Maximum 30 minutes (duration of the recovery phase)
  Time for the DROP index to reach 90% of its minimal value from the end of walking
Concordance of pain and ischemia during the treadmill test | Maximum 60 minutes (duration of each test)
  Observation of calf and non calf pain and calf and non-calf ischemia in patients reporting calf pain by history. Ischemia being defined as a minimal DROP value lower than minus 15 mmHg.
  Analysis of the concordance of localizations of pain and ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — UH in Angers (FRANCE)
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided
Data available under reasonable request